CLINICAL TRIAL: NCT06591806
Title: A Multicenter, Prospective, Longitudinal, Observational Study in Children and Adults With Stargardt Disease Related Atrophy Secondary to Biallelic Mutations in the ABCA4 Gene
Brief Title: An Observational Study in Children and Adults With Stargardt Disease
Status: Recruiting | Type: Observational
Sponsor: AAVantgarde Bio Srl (Industry)
Responsible Party: Sponsor
Other Study IDs: NHS-OBS-01
Record Dates: First submitted 2024-07-29; First posted 2024-09-19 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Stargardt Disease
Keywords: ABCA4
MeSH Terms: conditions — Stargardt Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This multicenter, prospective, longitudinal, observational study in approximately 80 subjects with Stargardt disease secondary to biallelic mutations in the ABCA4 gene (STGD1) aims to evaluate prognostic factors of disease progression, and to further characterize the patient population for future clinical studies.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects between 8 and 50 years of age at the time of enrolment.
2. Willingness to adhere to the protocol as evidenced by written informed consent if the subject is 18 years or older. If the subject is under 18 years of age, written assent must be obtained from the subject and written informed consent must be obtained from the subject's legally authorized representative (parent or legal guardian).
3. Confirmed mutation in the ABCA4 gene.

Exclusion Criteria:

1. History of uveitis.
2. Any ocular disease in either eye that may confound assessment of the retina morphologically and functionally.
3. Any pathology of the posterior segment other than ABCA4 retinopathy.
4. Presence of any other genetic mutation(s) that have been associated with retinal or macular dystrophy.

Ages: 8 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with Stargardt disease secondary to mutation in the ABCA4 gene
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
To measure the change from baseline in Fundus Autofluorescence | 24 months

CONTACTS AND LOCATIONS:
Locations (2):
- Retina Foundation of the Southwest, Dallas, Texas, United States
- Oslo University hospital Ullevål, Oslo, Norway